CLINICAL TRIAL: NCT05187975
Title: Integrated Rehabilitation in Treating Post-stroke Depression: Study Protocol for a Multicentre, Prospective, Randomised, Controlled Trial
Brief Title: Integrated Rehabilitation in Treating Post-stroke Depression
Acronym: IRTPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Third Affiliated hospital of Zhejiang Chinese Medical University (Other)
Collaborators: Zhejiang General Hospital of Armed Police (Other); Hangzhou Hospital of Traditional Chinese Medicine (Other); Jinhua Second Hospital (Unknown)
Responsible Party: Principal Investigator, Hong Gao, Deputy dean, The Third Affiliated hospital of Zhejiang Chinese Medical University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2021ZX010-B
Record Dates: First submitted 2021-12-03; First posted 2022-01-12 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Post-stroke Depression
Keywords: post-stroke depression; integrated rehabilitation; acupuncture; traditional Chinese medicine; repetitive transcranial magnetic stimulation; randomized controlled trial
MeSH Terms: interventions — Acupuncture Therapy; Medicine, Chinese Traditional; Transcranial Magnetic Stimulation; Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrated rehabilitation group (Experimental): This group will include 101 patients. On the basis of standard care, patients in this group will receive acupuncture, traditional Chinese medicine, repetitive transcranial magnetic stimulation .
  Interventions: Procedure: Acupuncture
- Standard care group (Active Comparator): The patients were recommended to take one oral tablet of paroxetine hydrochloride (20 mg) every morning after a meal for 4 weeks. Internal medicine includes lipid regulation, blood sugar control, anti-hypertension, anticoagulation, and other drugs. Moreover, general duty nursing and motor therapy are also needed.
  Interventions: Procedure: Acupuncture

INTERVENTIONS:
Procedure: Acupuncture — Acupuncture:
  Scalp acupuncture includes middle line of forehead (MS1), a front line by the forehead (MS2), and middle line of vertex (MS5), these acupoints are needled for 1 inch with the direction with scalp tilted 15-30 degrees.
  Body acupuncture includes Yintang (DU29), Taichong (LR3), Shenmen (HT7), Neiguan (PC6), Danzhong (RN17), Qimen (LR14), Taixi (KI3).
  Traditional Chinese medicine:
  Chaihushugan Power: Chaihu 12g, Chenpi 12g, Chuanxiong 9g, vinegar Xiangfu 9g, Zhike 9g, Shaoyao 9g, roasted Gancao 3g.
  Repetitive transcranial magnetic stimulation:
  The CCY-I magnetic field stimulator from Wuhan Irid Medical Equipment New Technology Co is used, with a frequency of 10Hz.
  Standard care:
  The same as the standard care group.
  Other Names: Traditional Chinese medicine; Repetitive transcranial magnetic stimulation; Standard care

SUMMARY:
Post-stroke depression (PSD) is a common complication of stroke that leads to dysfunction and reduces the quality of life. PSD exacerbates cognitive dysfunction, delays the recovery process, and increases the disability, mortality and recurrence rates of stroke. Therefore, early clinical treatments for PSD are important to improve the prognosis and restore the social functions of stroke patients.

Integrated rehabilitation has significant advantages in the treatment of PSD. First of all, there is a wide range of rehabilitation methods, such as acupuncture, traditional Chinese medicine, and repetitive transcranial magnetic stimulation, which have been proved to be effective for PSD. However, as the application of integrated rehabilitation becomes more and more widespread, its shortcomings are gradually emerging. For example, most of the treatment protocols used in clinical studies are based on personal experience of the investigators, a unified protocol has not yet been formed; treatment methods are still insufficient in standardization and reproducibility. More studies focus solely on the improvement of a certain symptom by a certain rehabilitation therapy, but ignore the important theoretical basis of the "holistic concept", thus showing the uneven clinical efficacy. For the above existing problems, it is necessary to conduct original and innovative research.

DETAILED DESCRIPTION:
This randomized controlled trial will enroll 202 PSD patients from the Third Affiliated Hospital of Zhejiang Chinese Medical University, Zhejiang General Hospital of Armed Police, Hangzhou TCM Hospital Affiliated to Zhejiang Chinese Medical University, and Jinhua Second Hospital. All patients will be randomly assigned to either the integrated rehabilitation group or the standard care group through a randomization system. The primary outcome will be assessed by hamilton depression (HAMD) scale, self-rating depression scale (SDS), and activity of daily living (ADL) scale. Secondary outcomes will include montreal cognitive assessment (MoCA) scale, the simple fugl-meyer assessment of motor function (FMA) scale and pittsburgh sleep quality index (PSQI).

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria of cerebral infarction or cerebral hemorrhage with depression disorder, the type of depression and the clinical syndrome of liver qi stagnation;
* Patients with clear consciousness, stable vital signs, ability to understand and cooperate with instructions, barthel index (BI) > 20, FMA (0-95), Mini-mental State Examination (MMSE) meet the following criteria: illiterate > 17, primary school level > 20, secondary school level (including technical secondary school) > 22, and college level (including junior college) > 23 points;
* 25 <= age <= 85 years, male or female;
* First episode of stroke, no personal or family history of mental disability before the stroke;
* Depression level as mild or moderate (HAMD scores >= 7 and <= 24);
* Depression symptoms occur after the stroke in a clear temporal sequence;
* The course of the PSD is limited to 2 weeks to 36 months after the stroke;
* Participants can understand the study protocol and written informed consent is signed.

Exclusion Criteria:

* Patients with acute brain trauma, brain infection, effusion, or tumor occupation;
* There are intracranial metals and other foreign bodies (such as orthopedic materials, arterial clips, etc.), cardiac pacemakers, deep brain stimulators, and other electronic devices;
* Previous seizures, including primary and secondary seizures；
* Patients have severe complications in cardiovascular, liver, kidney or psychiatric history ;
* There is a significant cognitive impairment (MMSE: literacy <= 17, primary school level <= 20, secondary school level (including technical secondary school) <= 22, and college level (including junior college) <= 23 points) or hearing impairment, aphasia;
* Coma, dying or chronic illness;
* Patients have taken psychotropic drugs or been treated for depression for nearly a month;
* People with unstable vital signs or patients with other mental disorders.

Ages: 25 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Estimated)
Dates: Start 2022-01-24 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in hamilton depression (HAMD) scale | Baseline, at 4-week during treatment, at 8-week follow-up
  Based on this large study of psychiatric outpatients with major depressive disorder we recommend the following severity ranges for the HAMD: no depression (0-7); mild depression (8-16); moderate depression (17-23); and severe depression (≥24). Severity classification on the Hamilton Depression Rating Scale J Affect Disord.
Change in self-rating depression scale (SDS) | Baseline, at 4-week during treatment, at 8-week follow-up
  Self-Rating Depression Scale (SDS) Description. This self-report scale was designed to quantify the severity of current major depression in 20 items. The scale was tested for psychometric properties. Various studies showed good to adequate results for validity.
Change in activity of daily living (ADL) scale | Baseline, at 4-week during treatment, at 8-week follow-up
  The Activities of Daily Living are a series of basic activities necessary for independent living at home or in the community. They are performed on a daily basis. There are many variations on the definition of the ADLs, but most organizations agree there are 5 basic categories.
  The Activities of Daily Living are a series of basic activities necessary for independent living at home or in the community. They are performed on a daily basis. There are many variations on the definition of the ADLs, but most organizations agree there are 5 basic categories.

SECONDARY OUTCOMES:
Change in montreal cognitive assessment (MoCA) scale | Baseline, at 4-week during treatment, at 8-week follow-up
  Montreal Cognitive Assessment scoring is based on a 30-point scale, with points awarded differently depending on the type of question asked. For instance, you can earn one point for each animal you identify in a picture, but listing the names of 13 fruits in under a minute gains you only two points.
Change in the simple fugl-meyer assessment of motor function (FMA) scale | Baseline, at 4-week during treatment, at 8-week follow-up
  Scoring is based on direct observation of performance. Scale items are scored on the basis of ability to complete the item using a 3-point ordinal scale where 0=cannot perform, 1=performs partially and 2=performs fully. The total possible scale score is 226.
  Points are divided among the domains as follows:
  Motor score: ranges from 0 (hemiplegia) to 100 points (normal motor performance). Divided into 66 points for upper extremity and 34 points for the lower extremity.
  Sensation: ranges from 0 to 24 points. Divided into 8 points for light touch and 16 points for position sense.
  Balance: ranges from 0 to 14 points. Divided into 6 points for sitting and 8 points for standing.
  Joint range of motion: ranges from 0 to 44 points. Joint pain: ranges from 0 to 44 points.
Change in pittsburgh sleep quality index (PSQI) | Baseline, at 4-week during treatment, at 8-week follow-up
  The range of values for questions 5 through 10 are all 0 to 3. Questions 1 through 9 are not allowed to be missing except as noted below. If these questions are missing then any scores calculated using missing questions are also missing. Thus it is important to make sure that all questions 1 through 9 have been answered.
  In the event that a range is given for an answer (for example, '30 to 60' is written as the answer to Q2, minutes to fall asleep), split the difference and enter 45.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Gao, Principal Investigator — Third Affiliated Hospital of Zhejiang Chinese Medical University
Locations (1):
- the Third Affiliated Hospital of Zhejiang Chinese Medical University, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Chen J, Shen K, Fan L, Hu H, Li T, Zhang Y, Gao H. Integrative medicine in treating post-stroke depression: Study protocol for a multicenter, prospective, randomized, controlled trial. Front Psychol. 2022 Aug 29;13:923506. doi: 10.3389/fpsyg.2022.923506. eCollection 2022. PMID 36110277